CLINICAL TRIAL: NCT01679782
Title: Phase 1 Impact of Nocturnal Desaturations on Central Motor Drive in COPD Patients: A New Insight on the Systemic Effects of the Disease.
Brief Title: Involvement of Nervous System in Muscle Weakness in COPD Patients
Acronym: DesCoM-1
Status: Completed | Type: Observational
Sponsor: 5 Santé (Other)
Collaborators: M2H laboratory, Montpellier University (Other); ANRT, National French Agency for Technological Researches (Unknown)
Responsible Party: Sponsor
Other Study IDs: FVIE_FA1
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, nervous system, peripheral muscle dysfunction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- COPD nocturnal desaturator: COPD patients who spend 30% of the nigth with a SaO2 < 90%.
- COPD no nocturnal desaturator: COPD patients who spend less than 30% of the night with a SaO2 < 90%
- control group: healthy sedentary subjects

SUMMARY:
The purpose of this study is to determine whether nervous system alterations and motor drive failure can contribute to muscle weakness in COPD during voluntary movement. If necessary, we will look after the role of nocturnal hypoxia in these alterations.

DETAILED DESCRIPTION:
COPD is a common disease that induces many systemic repercussions. Among these, peripheral muscle dysfunction is particularly deleterious because it leads to the decreases of the level of activity and the quality of life for patients. Movement involves activation of many structures, from the instructor, i.e. the brain, to the effector, i.e. the muscle. Netherless, the studies which have described peripheral muscle dysfunction have been focused on the muscle, so they have proposed a reducing vision of the phenomenon. Other studies have reported cerebral alterations in COPD, like cognitive disturbance, increase of the neuronal conduction time, and decrease of the white matter density, and were associated with chronic hypoxemia. Such alterations are consistent with the existence of a decrease of the central motor drive during voluntary movement in COPD patients. Therefore the study will aim to determine precisely which mechanisms are involved in peripheral muscle dysfunction in copd.

ELIGIBILITY:
Inclusion Criteria:

* COPD Patients at stage 2 and 3
* Healthy sedentary subjects

Exclusion Criteria:

* Epilepsy, pace-maker, nervous disorders

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of COPD patients and one group with healthy sedentary subjects
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Level of voluntary activation | 2h

CONTACTS AND LOCATIONS:
Overall Officials: Alain AV Varray, Pr, Study Director — M2H laboratory, Montpellier
Locations (1):
- Clinique du Souffle La Vallonie, Lodève, France

REFERENCES:
- [Derived] Alexandre F, Heraud N, Sanchez AM, Tremey E, Oliver N, Guerin P, Varray A. Brain Damage and Motor Cortex Impairment in Chronic Obstructive Pulmonary Disease: Implication of Nonrapid Eye Movement Sleep Desaturation. Sleep. 2016 Feb 1;39(2):327-35. doi: 10.5665/sleep.5438. PMID 26446126